CLINICAL TRIAL: NCT04467970
Title: Unicompartmental Knee Arthroplasty vs High Tibial Osteotomy: A Randomized Controlled Trial
Brief Title: Unicompartmental Knee Arthroplasty vs High Tibial Osteotomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Anter Ali Abdelhameed, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKAVSHTOARCT
Record Dates: First submitted 2020-07-06; First posted 2020-07-13 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis; Knee Arthroplasty
Keywords: Unicompartmental knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unicompartmental Knee Replacement (Experimental)
  Interventions: Procedure: Unicompartmental Knee Replacement
- High Tibial Osteotomy (Experimental)
  Interventions: Procedure: High Tibial Osteotomy

INTERVENTIONS:
Procedure: Unicompartmental Knee Replacement — Unicompartmental Knee Replacement involves replacement of the medial compartment of the knee in patients with anteromedial osteoarthritis.
  Arms: Unicompartmental Knee Replacement
Procedure: High Tibial Osteotomy — High Tibial Osteotomy involves medial wedge opening high tibial osteotomy in cases of anteromedial osteoarthritis.
  Arms: High Tibial Osteotomy

SUMMARY:
Valgus high tibial osteotomy (HTO) and unicompartmental knee arthroplasty (UKA) are established treatment options for patients with medial compartmental osteoarthritis (OA) of the knee.However, the clinical outcomes of these treatment modalities for unicompartmental OA have become subjects of debate.

DETAILED DESCRIPTION:
Although HTO for the correction of malalignment in the medial osteoarthritic knee has been shown to provide successful outcomes in some studies, it is technically difficult to achieve the ideal valgus position postoperatively, and the likelihood of postoperative complications after HTO is greater than that after UKA . As compared with HTO, UKA has been reported to provide better long-term results, to have a shorter time to full weight bearing, to allow easier rehabilitation, and to have fewer perioperative complications. Furthermore, indications for UKA are broadening, including younger and more active patients, since encouraging midterm and long-term results were published.

ELIGIBILITY:
Inclusion Criteria:

1. - Medial compartment osteoarthritis with exposed bone on both femur and tibia.
2. -Functionally intact Anterior Cruciate Ligament (superficial damage or splitting is acceptable)
3. -Full thickness and good quality lateral cartilage present
4. -Correctable intra-articular varus deformity (suggestive of functionally intact medical cruciate ligament) 5-Medically fit showing an American Society of Anesthesiologists (ASA) of 1 or 2

Exclusion Criteria:

1. Require revision knee replacement surgery.
2. Have rheumatoid arthritis or other inflammatory disorders.
3. Are unlikely to be able to perform required clinical assessment tasks.
4. Have symptomatic foot, hip or spinal pathology.
5. Previous knee surgery other than diagnostic arthroscopy and medial menisectomy.
6. Previously had septic arthritis.
7. Have significant damage to the patella-Femoral Joint especially on the lateral facet.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Pain and Function using Oxford Knee Score | at least two year follow up.
  this will be measured by using the Oxford Knee Score, a patient reported outcome questionnairewhich is A patient reported outcome measure highest score that could a patient get is 48 and means that good outcome and the lowest score to be obtained is 0 whick means poor outcome ( the higher the score,the better the outcome)

SECONDARY OUTCOMES:
Range of Motion and Function using the American Knee Society Score. | at least two year follow up
  this will be measured using the American Knee Society Score (AKSS). A clinician assessed score examining pain, stability, range of movement and function in which the maximum score to get is 100 and least score to get is 0 and the higher the score the better the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No